CLINICAL TRIAL: NCT03258008
Title: Phase II Trial of Utomilumab and ISA101b Vaccination in Patients With HPV-16-Positive Incurable Oropharyngeal Cancer
Brief Title: Utomilumab and ISA101b Vaccination in Patients With HPV-16-Positive Incurable Oropharyngeal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed the trial for infeasibility due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: ISA Pharmaceuticals B.V. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0145
Record Dates: First submitted 2017-08-21; First posted 2017-08-22 (Actual); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Malignant Neoplasms of Ill-defined Secondary and Unspecified Sites; Malignant Neoplasms of Lip Oral Cavity and Pharynx; Oropharyngeal Cancer
Keywords: Malignant neoplasms of lip oral cavity and pharynx; Malignant neoplasms of ill-defined secondary and unspecified sites; Oropharyngeal Cancer; Oropharyngeal squamous cell carcinoma; OPSCC; Human Papillomavirus - positive (HPV+); Utomilumab; PF-05082566; Anti-CD137; ISA101b
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Papillomavirus Infections | interventions — utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Utomilumab + ISA101b (Experimental): Utomilumab by vein every 4 weeks for up to 12 doses beginning on Cycle 1 Day 1.
  ISA101b as an injection under the skin every 4 weeks for 3 doses. Participants receive 2 injections each time.
  Interventions: Drug: Utomilumab; Biological: ISA101b

INTERVENTIONS:
Drug: Utomilumab — Utomilumab given by vein on Cycle 1 Day 1. Cycle 1-2 100 mg, Cycle 3-12 50 mg until progressive disease, toxicity, or 1 yr.
  Other Names: PF-05082566; Anti-CD137
Biological: ISA101b — ISA101b 100 mcg/peptide given subcutaneously every 4 weeks x 3 doses beginning cycle 1 day 1.

SUMMARY:
The goal of this clinical research study is to learn if utomilumab, when given with ISA101b, is able to shrink or slow the growth of tumors in patients with incurable HPV+ oropharyngeal squamous cell carcinoma.

This is an investigational study. Utomilumab and ISA101b are not FDA approved or commercially available. They are currently being used for research purposes only. The study doctor can explain how the study drugs are designed to work.

Up to 27 participants will be enrolled. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

There are 28 days in each study cycle.

You will receive utomilumab by vein every 4 weeks for up to 12 doses beginning on Cycle 1 Day 1. The drug will be given over about 1 hour each time you receive it.

You will receive ISA101b as an injection under the skin every 4 weeks for 3 doses. You will receive 2 injections each time. One may be in your arm and one in your leg.

Length of Study:

You may continue taking utomilumab for up to 1 year as long as your doctor thinks it is in your best interest. You will no longer be able to take the study drug(s) if intolerable side effects occur or if you are unable to follow study directions. You may not be able to take the study drug(s) if the disease gets worse, which is explained below.

Your participation on the study will be over after the follow-up visits.

Study Visits:

On Day 1 of Cycles 1-12:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be collected for routine tests, thyroid function tests, and liver function tests.
* If you can become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.
* During Cycles 1, 2, 3, 4, 8, and 12, blood (up to 10 tablespoons) will be drawn for biomarker testing (including genetic biomarkers).

At the end of Cycle 2 and every 8 weeks after that, you will have an MRI or CT scan to check the status of the disease.

Study Continuation:

If the disease appears to have gotten worse, you may still be eligible to continue receiving your assigned study drug(s). This is because you may be benefitting from the study drug(s) even though the tumor(s) got larger. Your doctor will discuss this with you.

If this happens, your doctor will talk to you about whether or not you want to continue. If you do continue taking part in the study, you will follow the study visits as described above.

However, there are risks of continuing to receive the study drug(s) because the disease may actually be getting worse. You are still at risk for side effects due to utomilumab and ISA101b. Continuing on this study could also delay starting other treatments. The disease may get worse to the point that you are no longer able to receive other treatments. There are also risks from the additional tests that may be performed, such as biopsies and blood draws. You and your doctor will discuss these possible risks, and you will be asked to decide if you want to continue receiving the study drug(s).

End-of-Treatment and Follow-up Visits:

At about 30 days after your last study drug dose:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be collected for routine tests, thyroid function tests, and liver function tests.
* If you are able to become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.

At about 70 days after your last study drug dose:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be collected for routine tests, thyroid function tests, and liver function tests.
* If you are able to become pregnant, blood (about ½ teaspoon) or urine will be collected for a pregnancy test.

You will also be called every 3 months up to 1½ years and asked about your health. Each call should last about 10-15 minutes.

If you stopped taking the study drug for reasons other than the disease getting worse, you will continue to have MRI/CT scans every 8 weeks. If the disease appears to get worse, or you start a new anticancer therapy, these scans will stop.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
2. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
3. Men and women >/= 18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 1.
5. Subjects with histologically- or cytologically-documented incurable Human Papillomavirus (HPV)-positive OPSCC. HPV-16 serotype will be assessed by Cervista assay.
6. Subjects can be treatment naïve or may have had two prior regimens for recurrent cancer. They must be naive to treatment with PD-1/L1 or CTLA-4 inhibitors.
7. Subjects must have progression within 6 months of platin exposure during definitive or palliative therapy.
8. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria; Radiographic Tumor Assessment performed within 28 days of study inclusion.
9. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site.
10. Subject entering the study will need to consent for mandatory biopsy at study entrance and as an optional procedure prior to C3 for biomarker evaluation. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is insufficient.
11. Prior chemotherapy, monoclonal antibody therapy, must have been completed at least 4 weeks prior to start. Radiotherapy or radiosurgery must have been completed at least 2 weeks prior to start.
12. All baseline laboratory requirements will be assessed and should be obtained within -14 days of study registration. Screening laboratory values must meet the following criteria i) White blood cells (WBCs) >/= 2000/microL ii) Neutrophils >/= 1500/microL iii) Platelets >/= 100 x 10^3/microL iv) Hemoglobin >/= 9.0 g/dL Patients must not be transfused for at least 14 days prior to study entry v) Serum creatinine of </=1.5 x upper limit of normal(ULN) or creatinine clearance(CrCl) > 50 mL/minute (using Cockcroft/Gault formula) Female CrCl= 0.85 x [(140 - age in years) x weight in kg]/(72 x serum creatinine in mg/dL) Male CrCl= 1.00 x [(140 - age in years) x weight in kg]/(72 x serum creatinine in mg/dL) vi) AST </= 2.5 x ULN vii) ALT </= 2.5 x ULN viii) Total bilirubin</= 1.5 x ULN (except subjects with Gilbert Syndrome who must have total bilirubin <3.0 mg/dl).
13. Women of childbearing potential (WOCBP) must use method(s) of contraception for 30 days + 5 half-lives (60 days) of the study drugs. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. Highly effective birth control in this study is defined as a double barrier method. Examples include a condom (with spermicide) in combination with a diaphragm, cervical cap, or intrauterine device (IUD). The individual methods of contraception should be determined in consultation with the investigator.
14. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
15. Women must not be breastfeeding.
16. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control for a period of 90 days plus the time required for the investigational drug to undergo 5 half- lives (60 days).

Exclusion Criteria:

1. Subjects with active CNS metastases are excluded. Subjects are eligible if CNS metastases are adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 4 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of </= 10 mg daily prednisone (or equivalent) for 2 weeks.
2. Subjects with carcinomatous meningitis.
3. Subjects with active, known or suspected systemic autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
5. Prior therapy with anti-CD137 or ISA101.
6. Subjects with a history of interstitial lung disease.
7. Other active malignancy requiring concurrent intervention.
8. Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
9. Subjects with toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue that have not resolved to grade 1 (NCI CTCAE version 4.03) or baseline before administration of study drug.
10. Subjects who have not recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment.
11. Treatment with any investigational agent within 28 days of first administration of study treatment.
12. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
13. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection.
14. History of allergy or intolerance (unacceptable adverse event) to study drugs components.
15. WOCBP who are pregnant or breastfeeding.
16. Women with a positive pregnancy test at enrollment or prior to administration of study medication.
17. Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results.
18. Prisoners or subjects who are involuntarily incarcerated.
19. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, BS,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 2018 to February 2019-Closed the trial for infeasibility due to slow accrual
Pre-assignment Details: 3 Participants registered to the trial, 1 was not eligible as screen fail.
Groups:
- Utomilumab and ISA101b: Treatment with Utomilumab every 4 weeks and 3 doses of ISA101b Vaccination for every 4 weeks first 3 cycles in Patients with HPV-16-Positive Incurable Oropharynx Cancer
Period: Overall Study
Arm/Group | Utomilumab and ISA101b
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who signed the consent are included in the baseline characteristics.
Arm/Group | Utomilumab and ISA101b
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Utomilumab Combined With ISA 101b in Patients With Incurable Human Papillomavirus - Positive (HPV+) Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: Overall Response Rate assessed by RECIST 1.1 Criteria
Time Frame: 9 weeks from start of treatment
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Utomilumab and ISA101b
Number analyzed (Participants) | 2
percentage of participants | 0 [0.0 to 0.8]

2. Secondary Outcome: Adverse Events of Utomilumab Combined With ISA 101b in Patients With Incurable Human Papillomavirus - Positive (HPV+) Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: Adverse events assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for grades 1-3.
Time Frame: Baseline, and continuously throughout the study at the beginning of each subsequent cycle up to 2 years
Measure: Number; unit: adverse events
Arm/Group | Utomilumab and ISA101b
Number analyzed (Participants) | 2
adverse events
  Grade 1 | 13
  Grade 2 | 0
  Grade 3 | 0

3. Secondary Outcome: Response Rate by irRC of Utomilumab Combined With ISA 101b in Patients With Incurable Human Papillomavirus - Positive (HPV+) Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: Response rate monitored by radiographic assessment.
Time Frame: Every-8-week schedule beginning from the first on-study assessment on Week 9 up to 2 years
Population: No data collected for Response Rate by irRC of Utomilumab Combined with ISA 101b in Patients with Incurable Human Papillomavirus - Positive (HPV+) Oropharyngeal Squamous Cell Carcinoma (OPSCC).
Arm/Group | Utomilumab and ISA101b
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival (PFS) of Utomilumab Combined With ISA 101b in Patients With Incurable Human Papillomavirus - Positive (HPV+) Oropharyngeal Squamous Cell Carcinoma (OPSCC)
Description: PFS defined as the time from first day of treatment to the date of the first documented tumor progression (per RECIST 1.1), or death due to any cause.
Time Frame: Every-8-week schedule beginning from the first on-study assessment on Week 9 up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Utomilumab and ISA101b
Number analyzed (Participants) | 2
months | 1.84 [1.84 to NA] — not estimable

ADVERSE EVENTS:
Time Frame: Adverse events will be captured from the time of the first protocol-specific intervention, until 30 days after the last dose of drug, unless the participant withdraws consent, through study completion an average of 24 months.
Arm/Group | Utomilumab and ISA101b
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Utomilumab and ISA101b (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Endocrine disorders - Other, specify Increased TSH Levels (Endocrine disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - Other, specify Rhinitis (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify pain at injection site (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03258008/Prot_SAP_000.pdf